## **Consent Form**

| I am father / mother of | | |
|---|---|---|
| program under the direction of A thorough description of the procedu | | understand that I may |
| withdraw my consent and discontinue | | |
| to me. | | |
| Date | Participant | |
| If illiterate A literate witness must sign (if possible, this person should be selected by the participant and should have no connection to the research team). Participants who are illiterate should include their thumb print as well. | | |
| I have witnessed the accurate reac<br>participant, and the individual has<br>individual has given consent freely. | had the opportunity to asl | <u>-</u> |
| Print name of witness | AND | Thumb print of |
| participant | | |
| Signature of witness | | |
| Date | | |
| Day/month/year | | |
| Statement by the researcher/person I have accurately read out the info and to the best of my ability made be done: | rmation sheet to the parer | |
| 1.<br>2. | | |
| 3. | | |
| I confirm that the parent was given<br>the questions asked by him/her hav<br>confirm that the individual has no<br>been given freely and voluntarily. | e been answered correctly | and to the best of my ability. I |
| Print Name of Researcher/person ta | aking the consent | |